CLINICAL TRIAL: NCT00631761
Title: Standardized Criteria to Judge Diagnostic Urethrocystoscopy Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Sam Siddighi, MD, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cystoscopy Project
Record Dates: First submitted 2008-02-27; First posted 2008-03-10 (Estimated); Last update posted 2008-08-19 (Estimated); Status verified 2008-08

CONDITIONS: Urethrocystoscopy Skills
Keywords: urethrocystoscopy; cystoscopy; objective structured assessment of surgical skills (OSATS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The intervention group will view a 20 minute video, receive a 30 minute didactic lecture on urethrocystoscopy, and 30 minute coaching/practice performing diagnostic cystoscopy on anatomic replicas of the human bladder.
  Interventions: Other: educational workshop
- 2 (Placebo Comparator): The control group will be instructed to read a urethrocystoscopy textbook chapter at home
  Interventions: Other: no intervention (usual resident activities)

INTERVENTIONS:
Other: educational workshop — The intervention group will view a 20 minute video, receive a 30 minute didactic lecture on urethrocystoscopy, and 30 minute coaching/practice performing diagnostic cystoscopy on anatomic replicas.
  Other Names: Objective structured assessment of surgical skills (OSATS), diagnostic cystoscopy,; urethrocystoscopy skills intervention, objective evaluation of procedure skills intervention,; educational workshops, cystoscopy classes, cystoscopy certificate
  Arms: 1
Other: no intervention (usual resident activities) — usual activities
  Arms: 2

SUMMARY:
Develop a tool to objectively quantify technical skills necessary to perform diagnostic cystoscopy (using Objective Structured Assessment of Technical Skills- OSATS).

Develop criteria by which surgeons skills in diagnostic cystoscopy can be evaluated or judged.

Develop an intervention (1.5 hour workshop) which can be replicated by other residency programs in order to enhance learning of diagnostic cystoscopy. The workshop should be adequate for practicing Gynecologists as well as they already have experience with diagnostic hysteroscopy which uses many of the same concepts.

DETAILED DESCRIPTION:
The OSATS and a written examination will be used to assess residents skills and knowledge pertinent to diagnostic urethrocystoscopy. All residents will be tested on anatomic replica of human bladder for baseline competency using the above tools. Then approximately half will be randomly selected to undergo an educational intervention (a workshop teaching diagnostic urethrocystoscopy). As we are interested in short-term acquisition, about a week later all residents will be retested using the same methods. Grades on the exam will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* All Obstetrics & Gynecology and Urology resident physicians training at the University of Cincinnati

Exclusion Criteria:

* Any above resident with extensive training in cystoscopy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
measure competency and change in urethrocystoscopy skills | 2 months

SECONDARY OUTCOMES:
Establish validity and reliability of measurement tools (OSATS) used to evaluate urethrocystoscopy skills | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sam Siddighi, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnat, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Siddighi S, Kleeman SD, Baggish MS, Rooney CM, Pauls RN, Karram MM. Effects of an educational workshop on performance of fourth-degree perineal laceration repair. Obstet Gynecol. 2007 Feb;109(2 Pt 1):289-94. doi: 10.1097/01.AOG.0000251499.18394.9f. PMID 17267826